CLINICAL TRIAL: NCT07067879
Title: The Effectiveness of a Novel Lip Product Containing Caulerpa Lentillifera Extract for Reducing Lip Hyperpigmentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREC-DCU2025-037
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Hyperpigmentation
Keywords: Lip hyperpigmentation; Seaweed; Antera3D; Lip care
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lip product application group (Experimental)
  Interventions: Other: Lip product

INTERVENTIONS:
Other: Lip product — Lip product containing Caulerpa lentillifera extract

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of the novel lip product containing Caulerpa lentillifera extract on the appearance and perception of dark lips in Thai adults aged 18 to 60 who report concerns about darkened lips. The main question it aims to answer is: Can the novel lip product containing C. lentillifera extract will significantly improve the appearance and perception of dark lips in Thai adults by reducing hyperpigmentation compared to baseline measurements?

Participants will apply the lip product twice a day, in the morning after breakfast and before bedtime, and refrain from using other lip products throughout the clinical trial period (7 days).

Researchers will compare the result to baseline measurements

ELIGIBILITY:
Inclusion Criteria:

* Understand the study protocol and provide informed consent after being informed of potential risks and benefits.
* Refrain from using any other lip products, including lipstick, lip gloss, or lip conditioners, during the study period.

Exclusion Criteria:

* Have a known allergy or sensitivity to cosmetic products or Caulerpa lentillifera.
* Are on medication one month prior to study commencement.
* Exhibit lip abnormalities such as malformation, inflammation, swelling, or sores.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-23 (Estimated); Primary Completion 2025-08-13 (Estimated); Study Completion 2025-08-13 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in improving lip hyperpigmentation | Baseline and 7 days
  Lip hyperpigmentation is assessed using Antera3D at baseline and 7 day after usage

SECONDARY OUTCOMES:
Change from baseline in improving lip dryness | Baseline and 7 days
  Lip dryness is assessed using Fotofinder system at baseline and 7 day after usage
Subjective assessment by participants | Baseline, day 1, and day 7
  Participants' evaluations will be collected through an online self-reported questionnaire. Subjective perceptions of lip color and dryness will be assessed using a 0-10 numerical darkness and dryness scale. Additionally, a satisfaction rating questionnaire will be administered to assess participant satisfaction with their lip appearance and the lip product on day 1 and day 7. The questionnaire will evaluate six key aspects of product performance;
  1. Overall satisfaction
  2. Effectiveness in hydration and moisturization
  3. Improvement in lip color and texture
  4. Ease of use and packaging design
  5. Sensory attributes such as texture and scent
  6. Occurrence of any adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Chulalongkorn university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No